CLINICAL TRIAL: NCT01659840
Title: Efficacy of Red and Infrared Lasers in Treatment of Temporomandibular Disorders - A Double-blind, Randomized, Parallel Clinical Trial
Brief Title: Efficacy of Red and Infrared Lasers in Treatment of Temporomandibular Disorders
Acronym: TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Olga Flecha, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: senhaodf
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Temporomandibular Disorders
Keywords: laser,; quality of life,; orofacial pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red laser (Other): On the pain points of muscle, laser was applied (8J/cm ²) with an interval of 48 hours between applications. In the joints with sensitivity, a dose of 4J/cm2 laser was applied with an interval of 48 hours between applications.
  Interventions: Radiation: Red laser
- Infrared laser (Other): On the pain points of muscle, laser was applied (8J/cm ²) with an interval of 48 hours between applications. In the joints with sensitivity, a dose of 4J/cm2 laser was applied with an interval of 48 hours between applications.
  Interventions: Radiation: Infrared laser

INTERVENTIONS:
Radiation: Red laser — On the pain points of muscle, laser was applied (8J/cm ²) with an interval of 48 hours between applications. In the joints with sensitivity, a dose of 4J/cm2 laser was applied with an interval of 48 hours between applications.
  Arms: Red laser
Radiation: Infrared laser — On the pain points of muscle, laser was applied (8J/cm ²) with an interval of 48 hours between applications. In the joints with sensitivity, a dose of 4J/cm2 laser was applied with an interval of 48 hours between applications.
  Arms: Infrared laser

SUMMARY:
The study hypothesis was that the red (600nm) and infrared (800nm) laser therapy have the same efficacy in relieving pain and improving the quality of life of TMD patients

DETAILED DESCRIPTION:
The aim of the present study was to evaluate and compare the efficacy of red (600nm) and infrared (800nm) laser therapy in relieving pain and improving the quality of life of TMD patients.

ELIGIBILITY:
Inclusion Criteria:

* systemic health;
* Temporomandibular Disorder diagnosed by the Research Diagnostic Criteria for Temporomandibular Disorders questionnaire (RDC);
* pain score ≥ 5 on palpation according to a visual and numerical scale (VNS)

Exclusion Criteria:

* participants who made frequent use of analgesics, NSAIDs and antidepressants;
* patients with previously undergone TMD treatment, or suffered facial trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
pain points of muscle and articulation | 180 days

SECONDARY OUTCOMES:
Quality of life | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Olga D Flecha, Professor, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Periodontics Clinic, Department of Dentistry, Diamantina, Minas Gerais, Brazil